CLINICAL TRIAL: NCT01312194
Title: Periapical Healing After One or Two-visits to Endodontic Treatment in Adolescents Patients
Acronym: PHAP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Federal do Rio de Janeiro (Other)
Responsible Party: Principal Investigator, Patricia de Andrade Risso, PHD, Universidade Federal do Rio de Janeiro
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 08176567-9
Record Dates: First submitted 2011-03-09; First posted 2011-03-10 (Estimated); Last update posted 2012-09-18 (Estimated); Status verified 2012-09

CONDITIONS: Periapical Periodontitis
Keywords: Periapical Periodontitis; Dental Pulp Necrosis; Root canal Therapy; Adolescent
MeSH Terms: conditions — Periapical Periodontitis; Dental Pulp Necrosis | interventions — Root Canal Therapy

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- One vist group (Experimental): All patients included in this treatment group will receive the complete endodontic treatment in a single visit.
  Interventions: Procedure: Root canal therapy in one visit
- Two-vist group (Active Comparator): All patients included in this treatment group will receive treatment in two visits. The first will be done chemo mechanical root canal preparation, the placement of the intracanal medication the basis of calcium hydroxide and coronal sealing. Ten to twelve days later, this medication is removed and the root canal will be permanently filled.
  Interventions: Procedure: Root Canal Therapy in two-vist

INTERVENTIONS:
Procedure: Root canal therapy in one visit — Patient was anesthetized with local anesthetic solutions, and the caries was removed. The tooth was isolated with rubber dam and access to pulp chamber was completed. Cleaning and shaping preparation was achieved with manual and rotatory endodontic instruments.The ideal working length was determined by an electronic apex locator and periapical radiography. Irrigation was performed with 5.25%NaOCl solution. The smear layer was removed by 10% citric acid. The cases were obturated with guta-percha cones using a lateral compaction filling technique as well as zinc oxide-eugenol-based root canal sealer. The teeth filled with a light-cured resin.
  Other Names: One visit root canal treatment; Single visit
  Arms: One vist group
Procedure: Root Canal Therapy in two-vist — The treatment protocol was the same as described for one visit group. In the first visit, after cleaning, shaping and smear layer removal, the root canals were medicated with a calcium hydroxide paste and sterile distilled water (1:1) and the pulp chamber was sealed with a minimum 3mm thickness temporary filling restoration. After 10-12 days, during the second visit, the medication was removed, and the cases were obturated with guta-percha cones using a lateral compaction filling technique as well as zinc oxide-eugenol-based root canal sealer. The teeth filled with a light-cured resin.
  Other Names: Multiple-visit of root canal treatment
  Arms: Two-vist group

SUMMARY:
The main objective of this study is the prevention and repair of apical periodontitis in lower molars with pulp necrosis after the execution of endodontic treatment in one or two visits in adolescent patients. Moreover, it is also observed the frequency of postoperative pain in endodontic treatment.

DETAILED DESCRIPTION:
This project is developed in adolescent patients who have need of endodontic treatment in necrotic molars. The patients were randomly divided into two groups of treatment: one and two visits. The treatment protocol is the same for both groups, except the number of visits and the use of intra canal medication in the group treated in two visits. Patients will be followed clinically and radiographically for a minimum period of two years. The data was collected by the evaluation of postoperative pain and to determine the healing of periapical lesions, characterizing the success of the treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Patients healthy
2. Not have taken analgesic, anti-inflammatory or antibiotic drugs during the 10 days prior to the beginning of treatment
3. Lower first or second permanent molars with complete root formation and dental pulp necrosis with or without symptoms

Exclusion Criteria:

1. Presence of periodontal diseases
2. Pulp calcification
3. Acute dent-alveolar abscesses
4. Hemorrhage in the canal after access

Ages: 11 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 120 (Actual)
Dates: Start 2004-05; Primary Completion 2007-05 (Actual); Study Completion 2008-08 (Actual)

PRIMARY OUTCOMES:
Healing Rate of one- versus two-visit endodontic treatment | Two years
  After completion of endodontic treatment in one or two visits, patients will be followed clinically and radiographically every 06 months for a minimum of two years to assess the prevention and repair of apical periodontitis.

SECONDARY OUTCOMES:
Postoperative pain of endodontic treatment | 60 days
  Following the completion of endodontic treatment in one or two visits, patients receive a clinical record for home monitoring of postoperative pain and return to clinic to conduct a follow-up clinical and radiographic. Pain is assessed using a numerical scale for pain.

CONTACTS AND LOCATIONS:
Overall Officials: Patrícia A Risso, Dentist, Principal Investigator — Universidade Federal do Rio de Janeiro; Antonio JL Cunha, doctor, Study Director — Universidade Federal do Rio de Janeiro
Locations (1):
- Federal University of Rio de Janeiro, Rio de Janeiro, Rio de Janeiro, Brazil

REFERENCES:
- [Result] Risso PA, Cunha AJ, Araujo MC, Luiz RR. Postobturation pain and associated factors in adolescent patients undergoing one- and two-visit root canal treatment. J Dent. 2008 Nov;36(11):928-34. doi: 10.1016/j.jdent.2008.07.006. Epub 2008 Sep 3. PMID 18771838
- [Result] de Andrade Risso P, da Cunha AJ, de Araujo MC, Luiz RR. Postoperative pain and associated factors in adolescent patients undergoing two-visit root canal therapy. Aust Endod J. 2009 Aug;35(2):89-92. doi: 10.1111/j.1747-4477.2008.00134.x. PMID 19703082